CLINICAL TRIAL: NCT00541684
Title: A Randomized, Double-Blind, Two Arm, Parallel Group Health Assessment Study of Losartan or Atenolol in Patients With Mild to Moderate Hypertension
Brief Title: Health Assessment Study (0954-946)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-946; 2007_624
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Duration of Therapy

INTERVENTIONS:
Drug: MK0954, /Duration of Treatment : 16 Weeks
Drug: Comparator : atenolol /Duration of Treatment : 16 Weeks

SUMMARY:
The study will look at the effects of losartan or atenolol on frequency of sexual intercourse in subjects with newly diagnosed mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with mild to moderate hypertension\
* Married male in stable heterosexual relationship
* No prior history of sexual dysfunction
* Satisfied with overall sex life
* Patient's spouse is in close proximity for the study
* Has had at least 2 but not more than 10 sexual intercourse events during the 2 week period prior to study start
* Patient able to visit doctor in the morning of each scheduled visit
* Able to complete the self administered health assessment questionnaire

Exclusion Criteria:

* Hypertension due to cancer, history of heart or circulatory problems
* History of mental disorder that might impair sexual function
* History or presence of drug or alcohol abuse
* Prior surgery for erectile dysfunction or other urological procedure
* No penile implant or assist devices
* History of chronic liver disease, history of diabetes
* History of severe life-threatening diseases such as, cancer, AIDS or positive HIV test
* Subjects with only 1 kidney
* Mental handicap or legal incapacity

Ages: 40 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2001-07-11 (Actual); Primary Completion 2003-01-23 (Actual); Study Completion 2003-01-23 (Actual)

PRIMARY OUTCOMES:
number of sexual intercourse events in a 2-week period | 2 Weeks

SECONDARY OUTCOMES:
sexual functioning score and overall sexual satisfaction score after 16 weeks | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC